CLINICAL TRIAL: NCT05535166
Title: SJiMB21: Phase 2 Study of Molecular and Clinical Risk-Directed Therapy for Infants and Young Children With Newly Diagnosed Medulloblastoma
Brief Title: Molecular and Clinical Risk-Directed Therapy for Infants and Young Children With Newly Diagnosed Medulloblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJiMB21; NCI-2022-07099 (Registry Identifier: NCI Clinical Trial Registration Program); R21CA280187 (NIH)
Record Dates: First submitted 2022-08-23; First posted 2022-09-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Medulloblastoma
Keywords: SJiMB21; Brain Cancer; Brain Tumors in Children; Medulloblastoma Sonic Hedgehog subgroup 1; Medulloblastoma Sonic Hedgehog subgroup 2; Medulloblastoma Sonic Hedgehog subgroup 3; Medulloblastoma Sonic Hedgehog subgroup 4; Medulloblastoma Sonic Hedgehog-not otherwise specified; Medulloblastoma G3; Medulloblastoma G4; Medulloblastoma indeterminate; MLPNet; Neural Net Classification Pipeline; Non-WNT non-SHH medulloblastoma; Posterior fossa syndrome; St. Jude Brain Tumor Studies; Treatment for Brain Tumors in Infants and Young Children; Untreated Childhood Medulloblastoma
MeSH Terms: conditions — Medulloblastoma; Brain Neoplasms | interventions — Methotrexate; Cisplatin; Vincristine; Cyclophosphamide; Carboplatin; Topotecan; Etoposide; pegfilgrastim; Filgrastim; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Stratum S-2 (Experimental): Patients with Sonic Hedgehog subgroup 2 (SHH-2), 0-2.99 years, or M0 and 3-4.99 years, will receive systemic high-dose methotrexate (HD-MTX) and conventional chemotherapy.
  Interventions: Surgery, Methotrexate, Cisplatin, Vincristine, Cyclophosphamide, Carboplatin, Topotecan, Pegfilgrastim, Filgrastim
  Interventions: Procedure: Surgical resection; Drug: Methotrexate; Drug: Cisplatin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Topotecan; Drug: Pegfilgrastim; Drug: Filgrastim
- Stratum S-1 (Experimental): Patients with SHH-1, SHH-3, SHH-4, or SHH-Not otherwise specified (NOS), 0-2.99 years, will receive intraventricular methotrexate (IVT-MTX) in parallel with systemic HD-MTX and conventional chemotherapy.
  Interventions: Surgery, Methotrexate, Cisplatin, Vincristine, Cyclophosphamide, Carboplatin, Topotecan, Pegfilgrastim, Filgrastim
  Interventions: Procedure: Surgical resection; Procedure: Ommaya/VPS; Drug: Cisplatin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Topotecan; Drug: Pegfilgrastim; Drug: Filgrastim; Drug: Methotrexate
- Stratum N (Experimental): Patients with Medulloblastoma (MB) group 3 or group 4 (G3/G4) or MB [including Non-WNT non-SHH medulloblastoma (NWNS) NOS or otherwise indeterminate cases] (0-2.99 years) will receive systemic HD-MTX and conventional chemotherapy only for radiation delaying purposes. At 3 years of age, these patients will receive risk-stratified craniospinal irradiation (CSI).
  Interventions: Surgery, Methotrexate, Cisplatin, Vincristine, Cyclophosphamide, Carboplatin, Topotecan, Etoposide, Pegfilgrastim, Filgrastim, Radiation
  Interventions: Procedure: Surgical resection; Drug: Methotrexate; Drug: Cisplatin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Carboplatin; Drug: Topotecan; Drug: Etoposide; Drug: Pegfilgrastim; Drug: Filgrastim; Radiation: Irradiation
- Cognitive Study Group I (educational video and games) (Experimental): Educational video and games
  Interventions: Other: Educational and Media Intervention
- Cognitive Study Group II (standard-of-care control) (Active Comparator): Standard-of-care (SOC) followed by educational video and games
  Interventions: Other: SOC, Educational and Media Intervention

INTERVENTIONS:
Procedure: Surgical resection — All participants enrolled will undergo surgical resection prior to treatment. The maximal resection that can be achieved without undue risk to the patient will be attempted, with decisions about feasibility and extent of resection left to the discretion of the neurosurgeon. In instances where an STR is the best extent of resection achieved prior to start of therapy, a "second-look" surgery may be performed between cycles of chemotherapy after discussion with the principal investigator.
  Other Names: surgical management
  Arms: Stratum N; Stratum S-1; Stratum S-2
Procedure: Ommaya/VPS — All participants enrolled on S-1 will undergo
  Other Names: surgical management
  Arms: Stratum S-1
Drug: Methotrexate — Route of administration: Intravenously (IV)
  Other Names: MTX; amethopterin
  Arms: Stratum N; Stratum S-2
Drug: Cisplatin — Route of administration: Intravenously (IV)
  Other Names: CDDP; cis-DDP; Platinol-AQ®
  Arms: Stratum N; Stratum S-1; Stratum S-2
Drug: Vincristine — Route of administration: Intravenously (IV)
  Other Names: Oncovin®
  Arms: Stratum N; Stratum S-1; Stratum S-2
Drug: Cyclophosphamide — Route of administration: Intravenously (IV)
  Other Names: Cytoxan®
  Arms: Stratum N; Stratum S-1; Stratum S-2
Drug: Carboplatin — Route of administration: Intravenously (IV)
  Other Names: Paraplatin®
  Arms: Stratum N; Stratum S-1; Stratum S-2
Drug: Topotecan — Route of administration: Intravenously (IV)
  Other Names: Hycamtin®
  Arms: Stratum N; Stratum S-1; Stratum S-2
Drug: Etoposide — Route of administration: Intravenously (IV)
  Other Names: VP-16; Vepesid®
  Arms: Stratum N
Drug: Pegfilgrastim — Route of administration: subcutaneous (SQ)
  Other Names: Udenyca®
  Arms: Stratum N; Stratum S-1; Stratum S-2
Drug: Filgrastim — Route of administration: subcutaneous (SQ) or Intravenously (IV)
  Other Names: GCSF; Neupogen®
  Arms: Stratum N; Stratum S-1; Stratum S-2
Radiation: Irradiation — All participants in stratum N will undergo craniospinal irradiation (CSI) with boost to the primary tumor site once they reach 36 months of age. The dose given is based on the molecular risk group and disease response to chemotherapy as noted in the arm descriptions. The type of radiation used includes conformal radiation therapy (photons) or intensity modulated radiation therapy (IMRT) or proton beam therapy.
  Other Names: Radiotherapy
  Arms: Stratum N
Other: Educational and Media Intervention — Participants watch a 75-minute caregiver education video program and receive access to interactive games on a smartphone or tablet throughout the optional cognitive study.
  Arms: Cognitive Study Group I (educational video and games)
Other: SOC, Educational and Media Intervention — Standard-of-care (SOC) treatment during main cognitive study. After the one-year serial cognitive evaluation, participants will be offered participation in the cognitive study group I intervention.
  Arms: Cognitive Study Group II (standard-of-care control)
Drug: Methotrexate — Route of administration: Intravenously (IV) & Intra Ventricular (IVT)
  Other Names: MTX; amethopterin
  Arms: Stratum S-1

SUMMARY:
This is a multi-center, multinational phase 2 trial that aims to explore the use of molecular and clinical risk-directed therapy in treatment of children 0-4.99 years of age with newly diagnosed medulloblastoma.

DETAILED DESCRIPTION:
The objectives of this study are:

Primary Objectives

* To estimate the progression free survival of SHH-2 infant (0-2.99 years) and young child (3-4.99 years) medulloblastoma patients treated with systemic HD-MTX- based chemotherapy only.
* To estimate the progression free survival of SHH-1 infant (0-2.99 years) medulloblastoma patients treated with systemic HD-MTX-based chemotherapy augmented with IVT-MTX.
* To estimate the progression free survival of G3/G4 infant (0-2.99 years) medulloblastoma patients treated with systemic chemotherapy and delayed risk- adapted CSI augmented with carboplatin.
* To compare cognitive outcomes among infants (0-2.99 years) and young children (3-4.99 years) treated with systemic chemotherapy only to patients treated with systemic chemotherapy and intra-ventricular chemotherapy or delayed risk- adapted craniospinal irradiation.

Secondary Objectives

* To investigate change in neurocognitive performance among infants (0-2.99 years) and young children (3-4.99 years) treated for medulloblastoma, and examine the impact of demographic factors (e.g., age at treatment, gender, and socioeconomic status), disease-related factors (e.g., presence of hydrocephalus, posterior fossa syndrome) and variants of proposed treatment regimen (e.g., systemic chemotherapy with or without IVT-MTX, radiation dosimetry to key brain structures, treatment-related ototoxicity) on cognitive late effects.
* To investigate which familial factors (e.g., family cohesion, family coping with medical management, parent-child interaction style) and environmental factors (e.g., parental verbal abilities, home literacy, adherence with rehabilitative therapies, participation in early intervention, school advocacy) associate with socioeconomic status and examine the impact of these factors on cognitive late effects.
* To evaluate the feasibility and acceptability of a caregiver education program paired with interactive neurodevelopmental games used to improve parent-child interactions, cognitive and social-emotional functioning in infants undergoing treatment for medulloblastoma. (funded by NCI via the R21CA280187)
* To estimate the magnitude of change in parent-child interactions following participation in a caregiver education paired with interactive neurodevelopmental games. (funded by NCI via the R21CA280187)
* To estimate the magnitude of change in cognition and social-emotional development associated with a caregiver education program combined with interactive neurodevelopmental games. (funded by NCI via the R21CA280187)
* To determine the extent of inter- and intra-patient variability in the plasma pharmacokinetics of high-dose systemic methotrexate, cyclophosphamide, vincristine, and topotecan in infants and young children with medulloblastoma, to assess potential covariates to explain this variability, and to explore associations between clinical effects and methotrexate, cyclophosphamide, vincristine, and topotecan pharmacokinetics.
* To determine the extent of inter- and intra-patient pharmacokinetic variability of methotrexate in ventricular CSF after intraventricular methotrexate dose administration in infants with medulloblastoma, and to explore associations between methotrexate CSF pharmacokinetics and clinical effects.

All participants enrolled will be treated with systemic chemotherapy post-surgical resection of the tumor. Participants will be assigned to treatment strata based first on tumor molecular group and subgroup assignment [SHH (including SHH-1, SHH-2, SHH-3, SHH-4 and SHH-NOS), G3, G4, (including NWNS NOS, or indeterminate cases] and then by clinical risk stratification (age and metastatic state).

Infants and young children on Stratum S-2 and infants on Stratum S-1 will be treated with chemotherapy-only strategies.

* Stratum S-2:

Patients on S-2 will receive 8 courses of chemotherapy consisting of:

* 4 Course A (A1A2A3A4)
* 2 Course B (B1B2)
* 2 Course C (C1C2) Courses repeat every 28 days/4 weeks.
* Stratum S-1:

Patients on S-1 will receive the same systemic chemotherapy regimen as S-2, with the addition of intraventricular (IVT)- MTX, administered via Ommaya reservoir, with each systemic MTX infusion. Each S-1 patient is scheduled to receive 12 doses of IVT-MTX. Each patient on S-1 will also receive 8 courses of combination chemotherapy. (4 Course A with IVT, 2 Course B with IVT and 2 Course C). Courses repeat every 28 days/4 weeks.

* Stratum N:

Stratum N participants will be treated with post-surgery chemotherapy until 36-months-of age followed by radiation CSI with Boost. There is no defined maximum number of systemic chemotherapy courses in stratum N. The length of chemotherapy (number of courses) will depend on the patient's age at enrollment. The chemotherapy plan for stratum N is divided into 5 sub-cohorts:

* Age ≥34 months and < 36 months: 4 cycles - 2 cycles (A1A2) prior to radiation and 2 cycles (E1, E2) post-radiation
* Age: ≥32 to <34 months-old: 4 cycles (A1A2A3A4)
* Age: ≥30 to <32 months-old: 6 cycles (A1A2A3A4 B1B2)
* Age: ≥28 to <30-months-old: 8 cycles (A1A2A3A4 B1B2 C1C2)
* Age: < 28 months-old: 8 cycles + multiple cycles of Course D until 36 months old (A1A2A3A4 B1B2 C1C2 D1D2D3D4…)

Courses A, B, C and E repeat every 28 days/4 weeks and Course D repeats every 42 days.

Prior to radiation therapy, around when stratum N patients achieve 36 months of age, they will be re-stratified onto substratum N-1, N-2 or N-3 based on their response to chemotherapy.

Patients who receive less than or equal to 4 cycles of systemic chemotherapy prior to CSI regardless of their substratum assignment (N-1, N-2 or N-3) will have their radiation therapy augmented by IV carboplatin. Carboplatin will be given to each of these patients 1-4 hours before each radiation fraction is delivered.

Patients enrolled in stratum N who have received only 2 courses of pre-radiation chemotherapy will receive 2 additional courses of adjuvant chemotherapy after completing CSI . The adjuvant chemotherapy consists of Cisplatin, Cyclophosphamide, and Vincristine. Patients who receive equal to 4 courses of systemic chemotherapy prior to CSI will have their radiation therapy augmented by IV carboplatin. The patients receiving more than 4 courses of chemotherapy prior to radiation will not receive additional adjuvant chemotherapy after completing CSI.

Patients will be followed for 84 months following enrollment.

ELIGIBILITY:
Inclusion Criteria - Screening Phase (All Patients)

* Participants with presumptive/suspected newly diagnosed medulloblastoma.
* Participant meets one of the following criteria at the time of screening:

  * Age < 36 months OR Age ≥ 36 months and < 60 months with presumptive/suspected non-metastatic disease
* Participant must have adequate tumor tissue from primary tumor for central review of pathology and molecular classification by methylation and IHC
* Participant must be able to begin treatment as outlined in the protocol within 36 days of definitive surgery (day of surgery is Day 0). In case a second surgery is clinically indicated to remove the residual tumor prior to starting treatment, the second surgery will be considered as the definitive surgery (Day 0).
* Parent or legal guardian can understand and is willing to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria - Screening Phase

* Participants with other clinically significant medical disorders (i.e., serious infections or significant cardiac, pulmonary, hepatic, psychiatric, or other organ dysfunction) that could compromise their ability to tolerate protocol therapy or would interfere with the study procedure.

Inclusion Criteria - Study Enrollment (All Patients)

* Participant must be < 60 months of age at time of enrollment.

  * Note: Each treatment stratum has additional specific age requirements
* Participant must have confirmation of newly diagnosed medulloblastoma per Central Review:

  * Central review includes histopathology, IHC and St. Jude Clinical Genomic Methylation Profiling conducted on MLPNet. If tissue or the extracted DNA does not meet quality control criteria for methylation analysis or if methylation classifier is unable assign molecular group/subgroup within the assigned classifier (MLPNet) parameters, then IHC will be used to define molecular group of these cases. IHC cannot be used to determine molecular subgroup. Therefore, IHC defined SHH patients will be enrolled on Stratum S-1 under "SHH-NOS", and all NWNS and indeterminate molecular group will be enrolled on stratum N.
  * Note: Diagnosis of medulloblastoma, as well as group and subgroup assignment, will be done by central pathology review at St. Jude only. No outside testing is allowed for trial enrollment.
* Participant must have disease staged by MRI of the brain and spine and by cytologic examination of CSF* and be placed into the following categories:

  * M0: no evidence of metastatic disease.

    * must include a negative CSF cytology result
  * M1: Tumor cells found in the CSF but no other evidence of metastasis
  * M2: Intracranial tumor beyond the primary tumor site
  * M3: Metastatic disease in the spine
  * M4: Extraneural metastatic disease
  * *All participants are to undergo CSF cytologic examination regardless of presence or absence of gross metastatic disease unless procedure is medically contraindicated. CSF is to be obtained by lumbar puncture (LP) performed at least 10 days after surgery. If LP is medically contraindicated, ventricular CSF from a shunt or Ommaya reservoir may be used for staging but this is not the preferred option due to lower sensitivity. If LP is medically contraindicated and the patient doesn't have a shunt or reservoir for CSF sampling, the treating physician should reach out to PI or Co-PI regarding decision on enrollment to SJiMB21. The decision to enroll without CSF cytology will be made on case-by-case basis.
  * Note: Participants who have M2 disease and positive CSF will be assigned to M3.
  * Note: Participants will be assigned to the highest stage number for which they meet eligibility.
  * Note: Treatment stratums may have additional stage requirements.
* Patient must have received no previous radiotherapy, chemotherapy, or other brain tumor-directed therapy other than corticosteroid therapy and surgery.
* Participant must have a Lansky performance score of > 30 (except for patients with posterior fossa syndrome.
* Participant must have adequate organ function prior to study entry, as defined by:

  * Absolute neutrophil counts (ANC) >750/mm^3
  * Platelet count ≥ 50,000/mm^3 without support of a platelet transfusion within 7 days
  * Hemoglobin ≥8.0 g/dL (with or without support of a blood transfusion).
  * Normal liver function as defined by Alanine aminotransferase (ALT) concentration ≤ 3 x 45 U/L and total bilirubin ≤ 3 x 1.0.
* Adequate renal function as defined by a serum creatinine concentration:

  * Age - 0 to <1year; Maximum Serum Creatinine (mg/dl) - Male 0.5; Female 0.5
  * Age - 1 to < 2years; Maximum Serum Creatinine (mg/dl) - Male 0.6; Female 0.6
  * Age - 1 to < 2yearsr; Maximum Serum Creatinine (mg/dl) - Male 0.8; Female 0.8
* Participant's parent or legal guardian has the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

Inclusion Criteria - Stratum S-2

* Participant must have confirmed diagnosis of the following medulloblastoma molecular group and subgroup per Central Review.

  * Medulloblastoma SHH-2
* Participant must meet one of the following criteria at time of enrollment:

  * Age <36 months OR Age ≥ 36 months and < 60 months with non-metastatic disease (M0) Inclusion Criteria - Stratum S-1
* Participant must have confirmed diagnosis of one of the following medulloblastoma molecular subgroups per Central Review.

  * Medulloblastoma SHH-1
  * Medulloblastoma SHH-3
  * Medulloblastoma SHH-4
  * Medulloblastoma SHH-NOS

    * Includes medulloblastoma cases that could not be assigned to a molecular subgroup using the DNA methylation classifier, but which are in the SHH group and/or cases defined as SHH by IHC.
* Participant must be < 36 months of age at time of enrollment

  * Note: Patients who are < 36 months of age, regardless of metastatic status (M0/M+), are eligible for enrollment on stratum S-1.

Inclusion Criteria - Stratum N

* Participant must have confirmed diagnosis of one of the following medulloblastoma molecular subgroups per Central Review.

  * Medulloblastoma G3
  * Medulloblastoma G4
  * Medulloblastoma - Not classified into SHH (i.e., NWNS or indeterminate)

    * Includes medulloblastoma cases that could not be assigned to a molecular group using the DNA methylation classifier but which are in the NWNS class and/or defined as NWNS by IHC.
* Participant must be <36 months of age at time of enrollment
* All NWNS patients (M+ and M0) are eligible for enrollment in stratum N

Exclusion Criteria - All Patients

* CNS embryonal tumor other than medulloblastoma, for example, patients with diagnosis of Atypical Teratoid/Rhabdoid Tumor (ATRT), PNET, Pineoblastoma, Ependymoma, and ETMR are excluded.
* Participant with prior treatment for medulloblastoma, including:

  * Radiotherapy
  * Chemotherapy
  * Cancer directed immunotherapy
  * Targeted agents
  * NOTE: Corticosteroid therapy is acceptable; prior treatment with chemotherapy, immunotherapy or targeted agents for non-cancer directed indications are acceptable as long as these have been stopped at least 14 days prior to start of therapy or 2 half-lives from last dose. (i.e., methotrexate for juvenile rheumatoid arthritis, JAK inhibitor therapy for eczema, etc.)
* Participant who is actively receiving any other investigational agents.
* Participant with other clinically significant medical disorders (i.e., serious infections or significant cardiac, pulmonary, hepatic, psychiatric, or other organ dysfunction) that could compromise their ability to tolerate protocol therapy or would interfere with the study procedures or results.

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival of SHH-2 infant (0-2.99 years) and young child (3-4.99 years) medulloblastoma patients treated with systemic HD-MTX-based chemotherapy only. | Up to 7 years after enrollment with PFS estimation occurring 2 years after treatment initiation of last patient
  Progression free survival (PFS) will be measured from treatment initiation to the earliest of disease progression or death from any cause in stratum S-2 eligible M0 patients who receive at least 1 dose of the chemotherapy regimen. Patients who have not experienced one of these events will be censored at their last date of contact. The Kaplan-Meier estimate of PFS at two years will be computed. PFS will be compared to St. Jude historical cohorts using hazard ratios with 95% confidence intervals.
Progression free survival of SHH-1 infant (0-2.99 years) medulloblastoma patients treated with systemic HD-MTX-based chemotherapy augmented with IVT-MTX. | Up to 7 years after enrollment with PFS estimation occurring 2 years after treatment initiation of last patient
  Progression free survival (PFS) will be measured from treatment initiation to the earliest of disease progression or death from any cause in stratum S-1 eligible SHH-1 patients who receive at least 1 dose of the chemotherapy regimen. Patients who have not experienced one of these events will be censored at their last date of contact. The Kaplan-Meier estimate of PFS at two years will be computed. PFS will be compared to St. Jude historical cohorts using hazard ratios with 95% confidence intervals.
Progression free survival of G3/G4 infant (0-2.99 years) medulloblastoma patients treated with systemic chemotherapy and delayed risk-adapted CSI augmented with carboplatin. | Up to 7 years after enrollment with PFS estimation occurring 2 years after treatment initiation of last patient
  Progression free survival (PFS) will be measured from treatment initiation to the earliest of disease progression or death from any cause in stratum S-N eligible patients who receive at least 1 dose of the chemotherapy regimen. Patients who have not experienced one of these events will be censored at their last date of contact. The Kaplan-Meier estimate of PFS at two years will be computed. PFS will be compared to St. Jude historical cohorts using hazard ratios with 95% confidence intervals.
IQ among infants and young children treated with systemic chemotherapy only compared to patients treated with systemic chemotherapy and intra-ventricular chemotherapy or delayed risk-adapted craniospinal irradiation | Baseline through 5 years after enrollment
  Change from baseline over time in intellectual function (IQ) will be assessed using different instruments as age appropriate. IQ will be measured in children 0-3:6 years of age using Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4), in children 3.0-5.11 years of age using Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV), and in children 6-10 years of age using Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V). Longitudinal analyses will be conducted using mixed models.
Executive function among infants and young children treated with systemic chemotherapy only compared to patients treated with systemic chemotherapy and intra-ventricular chemotherapy or delayed risk-adapted craniospinal irradiation | Baseline through 5 years after enrollment
  Change from baseline over time in executive functions will be assessed using different instruments as age appropriate. The Behavior Rating Inventory of Executive Function [BRIEF-P (ages 2-5:11) and BRIEF-2 (ages 6-18)] will assess behavioral manifestations of executive function. Longitudinal analyses will be conducted using mixed models.
Health-related quality of life among infants and young children treated with systemic chemotherapy only compared to patients treated with systemic chemotherapy and intra-ventricular chemotherapy or delayed risk-adapted craniospinal irradiation | Baseline through 5 years after enrollment
  Changes from baseline over time in health-related quality of life will be assessed using the PedsQL (ages 2 and older). Longitudinal analyses will be conducted using mixed models.

SECONDARY OUTCOMES:
Change in IQ among infants (0-2.99 years) and young children (3-4.99 years) treated for medulloblastoma | Baseline through 5 years after enrollment
  IQ will be assessed using different instruments as age appropriate. IQ will be measured in children 0-3:6 years of age using Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4), in children 3.0-5.11 years of age using Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV), and in children 6-10 years of age using Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V). The multiple instruments will be combined across all ages into one measure of standardized Full-Scale IQ. A linear mixed-effects regression model will be used to examine changes in IQ from baseline over time as related to demographic (e.g., age at treatment, gender, and socioeconomic status), disease-related (e.g., presence of hydrocephalus, posterior fossa syndrome), and treatment (e.g., systemic chemotherapy with or without IVT-MTX, radiation dosimetry to key brain structures, treatment-related ototoxicity) factors.
Change in executive function among infants (0-2.99 years) and young children (3-4.99 years) treated for medulloblastoma | Baseline through 5 years after enrollment
  This will be assessed using different instruments as age appropriate (The Behavior Rating Inventory of Executive Function [BRIEF-P (ages 2-5:11) and BRIEF-2 (ages 6-10)] will assess behavioral manifestations of executive function. A linear mixed-effects regression model will be used to examine changes in executive function from baseline over time as related to demographic (e.g., age at treatment, gender, and socioeconomic status), disease-related (e.g., presence of hydrocephalus, posterior fossa syndrome), and treatment (e.g., systemic chemotherapy with or without IVT-MTX, radiation dosimetry to key brain structures, treatment-related ototoxicity) factors.
Change in health-related quality of life among infants (0-2.99 years) and young children (3-4.99 years) treated for medulloblastoma | Baseline through 5 years after enrollment
  Health-related quality of life will be assessed using the PedsQL (ages 2 and older). A linear mixed-effects regression model will be used to examine changes in health-related quality of life from baseline over time as related to demographic (e.g., age at treatment, gender, and socioeconomic status), disease-related (e.g., presence of hydrocephalus, posterior fossa syndrome), and treatment (e.g., systemic chemotherapy with or without IVT-MTX, radiation dosimetry to key brain structures, treatment-related ototoxicity) factors.
Association of familial factors and environmental factors with socioeconomic status | Baseline through 5 years after enrollment
  Socioeconomic status will be measured using the Barratt Simplified Measure of Social Status (BSMSS). Generalized linear models will be used to investigate the association of socioeconomic status with familial factors (e.g., family cohesion, family coping with medical management, parent-child interaction style) and environmental factors (e.g., parental verbal abilities, home literacy, adherence with rehabilitative therapies, participation in early intervention, school advocacy)
Association of familial factors and environmental factors with cognitive late effects. | Baseline through 5 years after enrollment
  Linear mixed-effects models will be used to examine changes from baseline over time in cognitive outcomes (as described above) with familiar and environmental factors (as described above).
Evaluate family interest in caregiver education combined with interactive neurodevelopmental games. | Baseline through 6 months after enrollment
  The neurocognitive intervention consists of the Working for Kids (WFK) education, which is designed to improve parent understanding of the importance of the early learning environment on brain development, and First Pathways Game (FPG), which are interactive neurodevelopmental games designed for parents to play with their children to strengthen brain pathways for specific skills including communication, problem-solving and social emotional skills, motor skills, math skills and early science learning. Family interest in this intervention will be measured by the proportion of families approached enrolling on study.
Evaluate intervention feasibility by measuring the rate of participants completing a caregiver education combined with interactive. neurodevelopmental games. | Baseline through 6 months after enrollment
  The neurocognitive intervention consists of the Working for Kids (WFK) education, which is designed to improve parent understanding of the importance of the early learning environment on brain development, and First Pathways Game (FPG), which is an interactive neurodevelopmental games designed for parents to play with their children to strengthen brain pathways for specific skills including communication, problem-solving and social emotional skills, motor skills, math skills and early science learning. Intervention feasibility will be measured by the proportion of randomized participants completing at least 10 neurodevelopmental games.
Evaluate the acceptability of a caregiver education combined with interactive neurodevelopmental games. | Baseline through 6 months after enrollment
  The neurocognitive intervention consists of the Working for Kids (WFK) education, which is designed to improve parent understanding of the importance of the early learning environment on brain development, and First Pathways Game (FPG), which is an interactive neurodevelopmental games designed for parents to play with their children to strengthen brain pathways for specific skills including communication, problem-solving and social emotional skills, motor skills, math skills and early science learning. Acceptability will be measured as the proportion of caregivers reporting benefit from the intervention participation on a satisfaction questionnaire.
Magnitude of change in cognition and social-emotional development associated with a caregiver education program combined with interactive neurodevelopmental games. | Baseline and 6 months after enrollment
  Mean six-month change from baseline in cognition and social-emotional development as measured by DAYC-2 (parent interview) will be computed for families randomized to the intervention (described above) and for families randomized to the standard care control group.
To characterize the plasma systemic clearance (CL) of cyclophosphamide (CTX) in infants and young children with medulloblastoma. | Day 9 of the first course of A, AIVT, B or BIVT therapy and Days 4 and 5 of course C or Days 2 and 3 of E.
  Drug plasma concentrations will be simultaneously analyzed with a population pharmacokinetic approach, which permits characterizing typical pharmacokinetics and interindividual variability within the population. We will use a similar approach to what we have used in our previously published manuscripts. Cyclophosphamide CL will be estimated based on serial samples acquired during therapy.
To characterize the area under the concentration-time curve (AUC0-24h) of carboxyethylphosphoramide (CEPM) in infants and young children with medulloblastoma receiving cyclophosphamide. | Day 9 of the first course of A, AIVT, B or BIVT therapy and Days 4 and 5 of course C or Days 2 and 3 of E.
  Carboxyethylphosphoramide will be included in above described population pharmacokinetic approach. Based on the results of the population pharmacokinetic analysis, the CEPM AUC0-24h can be calculated.
To characterize the area under the concentration-time curve (AUC0-24h) of 4-hydroxy-cyclophosphamide (4OHCTX) in infants and young children with medulloblastoma receiving cyclophosphamide. | Day 9 of the first course of A, AIVT, B or BIVT therapy and Days 4 and 5 of course C or Days 2 and 3 of E.
  In a similar manner to the CEPM AUC0-24h, the 4-hydroxy-cyclophosphamide area under the curve AUC0-24h can be estimated based on the results of the population pharmacokinetic analysis.
To assess potential covariates (e.g., demographics, clinical chemistry) explaining inter- and intra-patient variability in in the plasma systemic clearance (CL) of CTX in infants and young children with medulloblastoma receiving CTX. | Data for CTX from Day 9 of the first course of A, AIVT, B or BIVT therapy and Days 4 and 5 of course C or Days 2 and 3 of E.
  A covariate analysis will be performed to investigate potential associations between the CTX CL pharmacokinetic parameter (outcome measure) and demographics and clinical chemistry data (covariates). Continuous covariates will be implemented according to a power model scaled to the population median covariate value. Categorical covariates will be modeled using an exponential change due to the covariate value. Significant covariates will be selected by using a classic forward/backward stepwise approach, with criteria P values of 0.05 and 0.01 for the forward and backward steps, respectively. Wald tests will be also used to test whether covariates should be kept in the model (criteria p-value<0.05) to explain the inter- and intra-patient variability in CTX CL values in infants and young children with medulloblastoma receiving CTX.
To assess potential covariates (e.g., demographics, clinical chemistry) explaining inter- and intra-patient variability in CEPM AUC0-24h in infants and young children with medulloblastoma receiving CTX. | Data for CEPM from Day 9 of the first course of A, AIVT, B or BIVT therapy and Days 4 and 5 of course C or Days 2 and 3 of E.
  A covariate analysis will be performed to investigate potential associations between the CTX AUC pharmacokinetic parameter (outcome measure) and demographics and clinical chemistry data (covariates). Continuous covariates will be implemented according to a power model scaled to the population median covariate value. Categorical covariates will be modeled using an exponential change due to the covariate value. Significant covariates will be selected by using a classic forward/backward stepwise approach, with criteria P values of 0.05 and 0.01 for the forward and backward steps, respectively. Wald tests will be also used to test whether covariates should be kept in the model (criteria p-value<0.05) to explain the inter- and intra-patient variability in CEPM AUC values in infants and young children with medulloblastoma receiving CTX.
To assess potential covariates (e.g., demographics, clinical chemistry) explaining inter- and intra-patient variability in 4OHCTX AUC0-24h in infants and young children with medulloblastoma receiving CTX. | Data for 4OHCTX from Day 9 of the first course of A, AIVT, B or BIVT therapy and Days 4 and 5 of course C or Days 2 and 3 of E.
  A covariate analysis will be performed to investigate potential associations between the 4OHCTX AUC pharmacokinetic parameter (outcome measure) and demographics and clinical chemistry data (covariates). Continuous covariates will be implemented according to a power model scaled to the population median covariate value. Categorical covariates will be modeled using an exponential change due to the covariate value. Significant covariates will be selected by using a classic forward/backward stepwise approach, with criteria P values of 0.05 and 0.01 for the forward and backward steps, respectively. Wald tests will be also used to test whether covariates should be kept in the model (criteria p-value<0.05) to explain the inter- and intra-patient variability in 4OHCTX AUC values in infants and young children with medulloblastoma receiving CTX.
To characterize the plasma systemic clearance (CL) of vincristine (VCR) in infants and young children with medulloblastoma. | Beginning on Day 15 of the first course of A or AIVT and B or BIVT (or Day 8 of one course E).
  As with cyclophosphamide, the vincristine drug plasma concentrations will be analyzed with a population pharmacokinetic approach, which permits characterizing typical pharmacokinetics and interindividual variability within the population. Vincristine CL will be estimated based on serial samples acquired during therapy.
To assess potential covariates (e.g., demographics, clinical chemistry) explaining inter- and intra-patient variability in VCR PK parameter (CL) in infants and young children with medulloblastoma receiving VCR. | Beginning on Day 15 of the first course of A or AIVT and B or BIVT (or Day 8 of one course E).
  A covariate analysis will be performed to investigate potential associations between the VCR CL pharmacokinetic parameter (outcome measure) and demographics and clinical chemistry data (covariates). Continuous covariates will be implemented according to a power model scaled to the population median covariate value. Categorical covariates will be modeled using an exponential change due to the covariate value. Significant covariates will be selected by using a classic forward/backward stepwise approach, with criteria P values of 0.05 and 0.01 for the forward and backward steps, respectively. Wald tests will be also used to test whether covariates should be kept in the model (criteria p-value<0.05) to explain the inter- and intra-patient variability in VCR CL values in infants and young children with medulloblastoma receiving VCR.
To characterize the plasma systemic clearance (CL) of topotecan (TPT) in infants and young children with medulloblastoma. | All samples acquired during each course C for domestic patients and patients at St. Jude only.
  The topotecan drug plasma concentrations will be analyzed with a population pharmacokinetic approach, which permits characterizing typical pharmacokinetics and interindividual variability within the population. Topotecan CL will be estimated based on serial samples acquired during course C of therapy.
To assess potential covariates (e.g., demographics, clinical chemistry) explaining inter- and intra-patient variability in TPT PK parameter (CL) in infants and young children with medulloblastoma receiving TPT. | All samples acquired during each course C for domestic patients and patients at St. Jude, only.
  A covariate analysis will be performed to investigate potential associations between the TPT CL pharmacokinetic parameter (outcome measure) and demographics and clinical chemistry data (covariates). Also included in this analysis will be concomitant medications given at the same as topotecan (i.e., cyclophosphamide), as well as concomitant adjuvant drugs given within 48 hr of topotecan dose in at least 30% of patients included in the analysis. Continuous covariates will be implemented according to a power model scaled to the population median covariate value. Patient age will be tested according to a Hill equation to reflect potential maturation process. Categorical covariates will be modeled using an exponential change due to the covariate value. Significant covariates will be selected by using a classic forward/backward stepwise approach, and a covariate was considered significant at P<0.05 for the forward addition and at the 0.01 for the backward addition.
To characterize the plasma systemic methotrexate (MTX) clearance (CL) in infants and young children with medulloblastoma. | Day 1 of each course A, AIVT, B, and BIVT.
  Drug plasma concentrations will be simultaneously analyzed with a population pharmacokinetic approach, which permits characterizing typical pharmacokinetics and interindividual variability within the population. We will use a similar approach to what we have used in our previously published manuscripts. Methotrexate CL will be estimated based on serial samples acquired during the first day of each course of therapy.
To characterize the area under the concentration-time curve (AUC0-24h) of 7-hydroxymethotrexate (7OHMTX) in infants and young children with medulloblastoma receiving methotrexate. | Day 1 of each course A, AIVT, B, and BIVT.
  7-hydroxymethotrexate will be included in above described population pharmacokinetic approach. Based on the results of the population pharmacokinetic analysis, the 7OHMTX AUC0-24h will be calculated.
To assess potential covariates (e.g., demographics, clinical chemistry) explaining inter- and intra-patient variability in MTX PK parameter CL in infants and young children with medulloblastoma receiving MTX. | Day 1 of each course A, AIVT, B, and BIVT.
  A covariate analysis will be performed to investigate potential associations between the MTX pharmacokinetic parameter CL (outcome measure) and demographics and clinical chemistry data (covariates). Continuous covariates will be implemented according to a power model scaled to the population median covariate value. Categorical covariates will be modeled using an exponential change due to the covariate value. Significant covariates will be selected by using a classic forward/backward stepwise approach, with criteria P values of 0.05 and 0.01 for the forward and backward steps, respectively. Wald tests will be also used to test whether covariates should be kept in the model (criteria p-value<0.05) to explain the inter- and intra-patient variability in MTX CL values in infants and young children with medulloblastoma receiving MTX.
To assess potential covariates (e.g., demographics, clinical chemistry) explaining inter- and intra-patient variability in 7OHMTX PK parameter AUC0-24h in infants and young children with medulloblastoma receiving MTX. | Day 1 of each course A, AIVT, B, and BIVT.
  A covariate analysis will be performed to investigate potential associations between the MTX pharmacokinetic parameter AUC (outcome measure) and demographics and clinical chemistry data (covariates). Continuous covariates will be implemented according to a power model scaled to the population median covariate value. Categorical covariates will be modeled using an exponential change due to the covariate value. Significant covariates will be selected by using a classic forward/backward stepwise approach, with criteria P values of 0.05 and 0.01 for the forward and backward steps, respectively. Wald tests will be also used to test whether covariates should be kept in the model (criteria p-value<0.05) to explain the inter- and intra-patient variability in 7OHMTX AUC values in infants and young children with medulloblastoma receiving MTX.

CONTACTS AND LOCATIONS:
Overall Officials: Giles W. Robinson, MD, Principal Investigator — St. Jude Children's Research Hospital; Aditi Bagchi, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (10):
- United States (10):
  - Lucille Packard Children's Hospital Stanford, Palo Alto, California
  - Orlando Health Arnold Palmer Hospital for Children, Orlando, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - C.S. MOTT Children's Hospital, University of Michigan, Ann Arbor, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center/Harold C Simmons Comprehensive Cancer Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — http://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042...